CLINICAL TRIAL: NCT05967806
Title: An International, Non-randomised, Non-interventional, Multicentre Study to Identify and Characterise Patients With CKD and High Proteinuria for Possible Participation in Future Renal Clinical Studies.
Brief Title: A Study to Identify and Characterise Patients With Chronic Kidney Disease and Proteinuria
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D4325C00007
Record Dates: First submitted 2023-07-20; First posted 2023-08-01 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-02

CONDITIONS: Renal Disease
Keywords: High Proteinuria
MeSH Terms: conditions — Kidney Diseases | interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

INTERVENTIONS:
Procedure: assessment — 2 ml volume of blood withdrawal

SUMMARY:
The purpose of the D4325C00007 study is to identify and characterise patients with known or newly diagnosed CKD for possible participation in future renal clinical studies and to obtain an overview on current treatment choices for this patient group in different regions.

ELIGIBILITY:
Inclusion criteria:

1. Male or female aged ≥ 18 years at the time of signing the informed consent
2. Express interest to participate in a future CKD clinical study
3. eGFR ≥ 20 to < 90 mL/min/1.73 m2 (eGFRcr[AS], Section 8.2.1) (Delgado et al 2022, Inker et al. 2021)
4. UACR ≥ 700 mg/g or UPCR ≥ 1000 mg/g based on urine sample at time of screening visit
5. Receiving RAS inhibitor therapy (ACEi or ARB) that has been at stable dosing for at least 4 weeks. Exceptions from this requirement will be made for participants who are unable to tolerate RAS inhibitor therapy
6. Provision of signed and dated written informed consent before any study-specific procedures

Exclusion criteria:

1. Known NYHA class III or class IV Congestive Heart Failure at the time of enrolment
2. Known T1DM
3. Known history of any life-threatening cardiac dysrhythmia (continuous or paroxysmal)
4. Known history of solid organ transplantation
5. Known history or ongoing allergy/hypersensitivity, as judged by the investigator, to SGLT2i (eg, dapagliflozin, canagliflozin, empagliflozin) or endothelin receptor antagonists (eg, ambrisentan, atrasentan, bosentan)
6. Known blood-borne diseases such as specified in Appendix B (category A and B)
7. Known pregnancy at the time for the visit or have an intention to become pregnant
8. Lupus nephritis, anti-neutrophil cytoplasmic autoantibody vasculitis, minimal change disease, autosomal dominant polycystic kidney disease (polycystic kidney disease), Alport syndrome, patients on renal replacement therapy, or clinical nephrotic syndrome with problematic oedema

Ages: 18 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: <3000
Sampling Method: Probability Sample
Enrollment: 2575 (Actual)
Dates: Start 2023-07-31 (Actual); Primary Completion 2024-08-30 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
Number of patients with UACR>700mg/g or UPCR >1000mg/g and eGFR 20-90 mL/min/1.73 m2 | approximately 10 months
  Summary statistics

SECONDARY OUTCOMES:
Number and sort of antihypertensive drugs among patients in different geographical regions | approximately 10 months
  Use of medications

CONTACTS AND LOCATIONS:
Locations (80):
- United States (17):
  - Research Site, Huntsville, Alabama
  - Research Site, Bakersfield, California
  - Research Site, Chatsworth, California
  - Research Site, San Carlos, California
  - Research Site, South Gate, California
  - Research Site, Tarzana, California
  - Research Site, Victorville, California
  - Research Site, Jacksonville, Florida
  - Research Site, Miami, Florida
  - Research Site, Kinston, North Carolina
  - Research Site, New Bern, North Carolina
  - Research Site, Wilmington, North Carolina
  - Research Site, Winston-Salem, North Carolina
  - Research Site, Greenville, South Carolina
  - Research Site, Pearland, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Arlington, Virginia
- Argentina (2):
  - Research Site, Buenos Aires
  - Research Site, Santa Fe
- Brazil (4):
  - Research Site, Belém
  - Research Site, Botucatu
  - Research Site, São José do Rio Preto
  - Research Site, São Paulo
- Canada (2):
  - Research Site, London
  - Research Site, Waterloo
- China (9):
  - Research Site, Beijing
  - Research Site, Guangdong
  - Research Site, Hubei
  - Research Site, Hunan
  - Research Site, Jiangsu
  - Research Site, Shenzhen
  - Research Site, Sichuan
  - Research Site, Wenzhou
  - Research Site, Zhejiang
- India (3):
  - Research Site, Bangalore
  - Research Site, Delhi
  - Research Site, Nadiād
- Poland (6):
  - Research Site, Chrzanów
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Radom
  - Research Site, Rzeszów
  - Research Site, Warsaw
- Slovakia (6):
  - Research Site, Košice
  - Research Site, Lučenec
  - Research Site, Prešov
  - Research Site, Púchov
  - Research Site, Rožňava
  - Research Site, Trebišov
- South Africa (6):
  - Research Site, Benoni
  - Research Site, Chatsworth
  - Research Site, Durban
  - Research Site, Lenasia
  - Research Site, Parow
  - Research Site, Soweto
- Sweden (4):
  - Research Site, Linköping
  - Research Site, Rättvik
  - Research Site, Stockholm
  - Research Site, Uppsala
- Taiwan (6):
  - Research Site, Kaohsiung City
  - Research Site, New Taipei City
  - Research Site, Taichung
  - Research Site, Taipei
  - Research Site, Taoyuan District
  - Research Site, Yongkang District
- Thailand (4):
  - Research Site, Bangkok
  - Research Site, Chiang Mai
  - Research Site, Khon Kaen
  - Research Site, Songkhla
- Turkey (Türkiye) (8):
  - Research Site, Adapazarı
  - Research Site, Afyonkarahisar
  - Research Site, Ankara
  - Research Site, Antalya
  - Research Site, Bursa
  - Research Site, Kahramanmaraş
  - Research Site, Kayseri
  - Research Site, Kocaeli
- Vietnam (3):
  - Research Site, Haiphong
  - Research Site, Hà Nội
  - Research Site, Ho Chi Minh City

REFERENCES:
- See also: D4325C00007_redacted CSR synopsis-exploratory-study-report-abbreviated_redacted — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D4325C00007&attachmentIdentifier=08d7287e-2b35-4290-a02b-5b1939da5bc4&fileName=D4325C00007_redacted_CSR_synopsis-exploratory-study-report-abbreviated.pdf&versionIdentifier=